CLINICAL TRIAL: NCT06209086
Title: Evaluation of the Dentoskeletal Effects of Skeletal Anchored Versus Incisal Capped Twin Block Appliance in the Treatment of Class II Malocclusion
Brief Title: Effects of Skeletal Anchored Versus Incisal Capped Twin Block Appliance in Class II Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Elabd, teaching assistant - orthodontic department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ortho
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- incisal capped twin block (Active Comparator): The incisal capped Twin Block, which was used for the first group composed of two parts. The upper part had labial bow over labial surface of upper anterior teeth using Adam and ball clasps for retention.
  The lower part included ball clasp between lower anterior teeth and Adam clasp on lower first premolar with the additional modifications:
  * The lower incisors were capped with acryl.
  * lower incisors were relieved from the lingual side with wax.
  Interventions: Device: skeletal anchored twin block
- skeletal anchored twin block (Active Comparator): This appliance was constructed as the modified Twin Block used for the incisal capped appliance in addition to the following modifications:
  * Addition of mini-implants interdentally between the mandibular second premolar and mandibular first molar.
  * Wire hooks: wire hook element in the lower part of the appliance was incorporated in the region of incisal capping with free end projecting at the canine region on both sides.
  * Intra-oral elastics were attached from the mini-implant to the wire hook bilaterally.
  Interventions: Device: skeletal anchored twin block

INTERVENTIONS:
Device: skeletal anchored twin block — This appliance was constructed as the modified Twin Block used for the first group in addition to the following modifications:
  * Addition of mini-implants interdentally between the mandibular second premolar and mandibular first molar.
  * Wire hooks: wire hook element in the lower part of the appliance was incorporated in the region of incisal capping with free end projecting at the canine region on both sides.
  * Intra-oral elastics were attached from the mini-implant to the wire hook bilaterally.

SUMMARY:
: the purpose of this study was to evaluate the dento-skeletal effects of the mini-implant supported Twin Block versus the incisal capped appliance in the treatment of skeletal class II patients with mandibular retrognathism.

Methods: Twenty patients with skeletal class II mandibular retrusion were included in the study. They were recruited with a random and equal allocation into 2 groups. The first group was treated with incisal capped TB without skeletal anchorage. The second group were treated with mini-implant supported TB. The mini-implants were inserted in the inter-radicular region between the mandibular second premolar and first molar. Intra-oral elastics were attached from the mini-implant to the wire hook in the canine region of the lower part of the TB and they were changed every 24 hrs. 100 to 150 gm of force was applied. Cephalometric radiographs were acquired at the beginning (T1) and end of treatment (T2). The paired-samples and independent-samples t-tests were used to evaluate and compare the changes within groups and between groups, respectively.

DETAILED DESCRIPTION:
Twenty patients with skeletal class II mandibular retrusion were included in the study. They were recruited with a random and equal allocation into 2 groups. The first group was treated with incisal capped TB without skeletal anchorage. The second group were treated with mini-implant supported TB

Appliance construction:

1. Bite registration

   * First, the administrator measured the overjet using calibrated poly gauge from the incisal edge of the most protruded upper incisor to the facial surface of the lower central incisor.
   * Then, a wax bite was done using the Exacto bite or Projet Bite Gauge (12) with the addition of softened horseshoe wafer of medium hard wax for easy registration of the bite. The mandible was anteriorly positioned to make an edge-to-edge relationship parallel to the functional occlusal plane. At the same time, the posterior vertical separation between arches was with an adequate width between 4-5 mm. The excess was removed along the gingiva, retromolar region and on the palatal tissue if found.
   * During bite registration, making sure the upper and lower mid lines of the patient were the same as in his original distal occlusion as long as there was no functional shift of the mandible.
2. Design of the appliance A-modified twin block The incisal capped Twin Block, which was used for the first group composed of two parts. The upper part had labial bow over labial surface of upper anterior teeth using Adam and ball clasps for retention.

The lower part included ball clasp between lower anterior teeth and Adam clasp on lower first premolar with the additional modifications:

* The lower incisors were capped with acryl.
* lower incisors were relieved from the lingual side with wax. B-Mini-implant supported modified Twin Block .

This appliance was constructed as the modified Twin Block used for the first group in addition to the following modifications:

* Addition of mini-implants interdentally between the mandibular second premolar and mandibular first molar.
* Wire hooks: wire hook element in the lower part of the appliance was incorporated in the region of incisal capping with free end projecting at the canine region on both sides.
* Intra-oral elastics were attached from the mini-implant to the wire hook bilaterally.

Insertion of the Mini-implants:

* Two orthodontic Dentaurum miniscrew (1,6*8 mm) were used in this study which were intended to be placed bilaterally on lower arch between the mandibular second premolar and first molar.
* Surgical mesh was used as a guide tool in the mouth for accurate placement of the mini- implants. The mesh guide was first adapted on the cast of each patient and it was extended from the mesial contact of the lower second premolar to the distal one of the first permanent molar and extended apically to the depth of the sulcus. Then it was tried in the patient mouth to avoid any extension that might cause injury to the oral mucosa of the patient.
* The mesh was then stabilized on the patient mouth by using rubber base impression material .
* Then peri apical radiographs were taken to use it as a guide for the precise placement of the mini-implant .
* The purpose of using rubber base material to ensure the accurate position of the mesh guide to be the same during the insertion of the mini screw intra orally.
* After locating the precise point of insertion of the mini-implant with the help of mesh guide and before the insertion of them, the mini-implants were self-drilled using a straight screwdriver in the attached gingiva at the mucogingival line leaving 0.5 mm of the transmucosal collar outside the mucosa. This amount of collar outside was planned to facilitate the insertion of intra oral elastics. The implants were inserted at approximately 20-30 degrees to the occlusal plane.
* Peri apical radiograph was then taken to the right and left sides to verify the position of mini-implant with the cone of the machine is directed perpendicular to the film .
* Intra oral elastics: elastics of dimension 3⁄8 (4 oz., 150 gm of force) was attached to the wire hooks to exert a class I distalizing force taking anchorage from mini-implants. The force is measured using Morelli force gauge.

Delivery of appliance and patient instruction:

The appliance was checked for fitting in the patient's mouth systemically, in the upper jaw then in the lower jaw separately and then the two parts were checked together when the jaws were closed. We checked the presence of any roughness, sharp areas or undercuts that may cause discomfort to the patients.

The patients and parents were instructed to:

* Put on the twin block appliance full time 24 hours a day.
* Maintain good oral hygiene, brush teeth and the appliance after each meal.
* Attain orthodontic clinic every three weeks.
* Change the elastics every 24 hour.
* Accordingly, at each appointment, the patient was checked for the outcomes of mandibular advancement and presence or absence of posterior cross-bite and subsequent need for opening of the expansion screw.
* At the time of activation, another registration wax bite was taken in this time for edge to edge upper and lower incisors.

Retention When the overjet was corrected; a retention appliance was constructed to correct lateral open bite that resulted from presence of occlusal bite blocks.

ELIGIBILITY:
Inclusion Criteria:

* early permanent dentition (ages 9 to 14)
* mandibular retrusion-related class II skeletal deformity
* overjet more than 4mm.

Exclusion Criteria:

* systemic diseases
* congenital craniofacial deformity
* cleft lip or palate
* unusual habits
* previous orthodontic treatment.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-19 (Actual)

PRIMARY OUTCOMES:
dentoskeletal effects of skeletal anchored versus incisal capped twin block appliance in the correction of skeletal class II malocclusion | 11 months
  the study include 20 patients with skeletal class II malocclusion who were treated with incisal capped and skeletal anchored twin block advancement of mandible with controlling the position of lower incisors in the second group

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa A Elabd, master, Principal Investigator — mansoura univeristy
Locations (1):
- Dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No